CLINICAL TRIAL: NCT05304286
Title: Psychophysical and Neural Mechanisms Contributing to Chronic Post-Surgical Pain in Adolescents and Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Christine B. Sieberg, PhD, Associate Professor of Psychology, Department of Psychiatry, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P000634
Record Dates: First submitted 2021-12-22; First posted 2022-03-31 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Chronic Post-surgical Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT Group Intervention (Active Comparator): We will evaluate the effects of an Acceptance and Commitment Therapy (ACT) one-day group intervention (with 1-month post group zoom booster session) on the functional near-infrared spectroscopy (fNIRS) signal in groups of adolescents and adult patients diagnosed with CPSP at >3 months post major orthopedic surgery.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Treatment as Usual (No Intervention): Treatment as Usual (TAU) for those with CPSP

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — The aim of ACT is to address avoidance behaviors by increasing openness to difficult experiences, such as pain, and to develop an awareness of behavioral options that will aid to facilitate behavior change processes that are in accord with living a values-based life.
  Arms: ACT Group Intervention

SUMMARY:
The current project will (1) enhance our understanding of the neurobiology of chronic post-surgical pain (CPSP); (2) provide a metric to follow patients with CPSP in the clinic; (3) provide a metric for those who will chronify; and (4) understand the age-related differences in CPSP. Ultimately, an improved comprehension of mechanisms linked to CPSP will provide finer tools for optimizing the selection of treatments for individual patients. Moreover, data that demonstrates the underlying pathobiological pain mechanism(s) active in CPSP, particularly those non-responsive to current therapies, may be used to validate novel strategies both pharmacological and non-pharmacological.

DETAILED DESCRIPTION:
In this mechanistic clinical trial, participants will be randomized into either a one-day (5 hours) group workshop based on Acceptance and Commitment Therapy (ACT) and a one-month post workshop zoom individual booster session or Treatment as Usual (TAU).

Dr. Sieberg will conduct the groups with assistance from the RA. Dr. Sieberg is a licensed clinical psychologist, who has delivered manualized ACT for chronic pain in her clinical practice. The intervention follows a manual patterned after an existing 1-day ACT intervention for chronic pain and will be adapted to meet the needs of patients with ongoing CPSP. Topics covered in the workshop include: (1) mindfulness of troublesome thoughts, feelings, and physical sensations; (2) willingness to face and accept experiences that cannot be changed; (3) identifying values; and (4) promoting behavior changes that support value-based action.

The goal of the ACT intervention is to increase awareness of thoughts, feelings, and behaviors that exacerbate pain while minimizing avoidance that interferes with engagement in valued action. Participants will also receive an individually tailored 30-minute booster session via zoom one month following the workshop. During the booster session, ACT principles will be reinforced and the participant will work together with Dr. Sieberg to problem-solve and address any difficulties engaging in ACT exercises and practices.

ELIGIBILITY:
Inclusion Criteria:

--Females and males aged 12 and older who have previously undergone surgery at least 6 months ago and have chronic post surgical pain (3 months after surgery or longer)

Exclusion Criteria:

* Inability to speak sufficient English or another language that can be interpreted orally and for questionnaires with the research team
* Severe cognitive impairment by history (e.g., intellectual disability, severe head injury)
* Patients with significant psychiatric disorders
* Use of illegal hard drugs including MDMA, heroin, methamphetimes, amphetamines, cocaine, ketamine, benzodiazepines, and phencyclidine. Absence of such drugs will be confirmed in a urine drug screen during the visit. If prescription medication includes any of these compounds, that medication is not exclusionary.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain acceptance using the Chronic Pain Acceptance Questionnaire - Revised (CPAQ-R) | 5 years
  The 20-item CPAQ-revised has been designed to measure acceptance of pain. The acceptance of chronic pain is thought to reduce unsuccessful attempts to avoid or control pain and thus focus on engaging in valued activities and pursuing meaningful goals. The items on the CPAQ are rated on a 7-point scale from 0 (never true) to 6 (always true). To score the CPAQ, add the items for Activity engagement and Pain willingness to obtain a score for each factor. To obtain the total score, add the scores for each factor together. Higher scores indicate higher levels of acceptance

SECONDARY OUTCOMES:
Functional brain metrics using fNIRS | 5 years
  To identify alterations in brain metrics and define changes in brain function as a correlate of pain, participants will undergo an fNIRS brain scan. The following regions of interest will be explored: primary somatosensory cortex (SI) and the medial prefrontal cortex (mPFC). fNIRS is a non-invasive neuroimaging method that employs near infrared light to measure cortical hemodynamic changes. The near infrared light penetrates the superficial layers (the skin and the skull) to then reach the cortex. Throughout the travel within the tissue, light is mostly absorbed by chromophores, namely the oxygenated hemoglobin (HbO) and deoxygenated hemoglobin (HbR).

CONTACTS AND LOCATIONS:
Overall Officials: Christine B. Sieberg, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No